CLINICAL TRIAL: NCT04050163
Title: Safety and Preliminary Efficacy Study of Intravenous Administration of MiSaver® (Myocardial Infarction Saver) After Acute Myocardial Infarction, a Phase I/IIa Clinical Trial.
Brief Title: MiSaver® Stem Cell Treatment for Heart Attack (Acute Myocardial Infarction)
Acronym: MiSaver®
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Honya Medical Inc (Industry)
Collaborators: Chung Shan Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: csho19052112001
Record Dates: First submitted 2019-08-06; First posted 2019-08-08 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Myocardial Infarction
Keywords: Heart Attack
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: Sequential dose escalating
Who Masked: Participant
Masking Description: Single/participant blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low Dose (Experimental): Cells dosage, 0.5x10^7 cells/kg body weight
  Interventions: Biological: MiSaver®
- Intermediate Dose (aka Effective or High) (Experimental): Cells dosage, 1.6x10^7 cells/kg body weight
  Interventions: Biological: MiSaver®
- Toxic Dose (Experimental): Cells dosage, 5.0 x10^7 cells/kg body weight
  Interventions: Biological: MiSaver®

INTERVENTIONS:
Biological: MiSaver® — Intravenous administration of MiSaver® Stem Cell via peripheral vein access.
  Other Names: stem cells

SUMMARY:
The objective of the present study is to establish the safety and efficacy of MiSaver® Stem Cell Treatment After a Heart Attack (Acute Myocardial Infarction)

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 20~80
* Acute Myocardial Infarction 1 to 10 days
* Cardiac enzyme CK-MB or Troponin > 2X of high-end normal value
* ST-elevation on EKG (STEMI)
* Presence of regional wall motion abnormality
* Left ventricular ejection fraction (LVEF) of ≤40%
* Hemodynamically stable past 24 hour
* Participants with adequate pulmonary function
* Peripheral artery oxygen saturation ≥97%
* Karnofsky performance status scores of ≥60.

Exclusion Criteria:

* Age <20 or >80
* Pregnant or breast feeding
* Positive adventitious infections (such as HIV, hepatitis )
* Revascularization via coronary artery bypass surgery is required
* Coronary revascularization procedures is anticipated during the 6-month study period
* Severe aortic or mitral valve narrowing
* Evidence of life-threatening arrhythmia on baseline electrocardiogram (ECG)
* Short of breath unable to receive PCI examination or treatment
* Malignant tumor
* Hematopoietic dysplasia
* Severe organ disease
* With less than 1 year of life expectancy
* Chronic kidney disease with CCr<20ml/min
* Kidney disease on renal dialysis

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-01-26 (Actual); Primary Completion 2023-05-04 (Actual); Study Completion 2023-05-04 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events | 12 months
  Number of Adverse Events

SECONDARY OUTCOMES:
Left ventricle stroke volume | 12 months
  Echocardiogram assessment on left ventricle stroke volume (volume of blood pumped from the left ventricle per beat (ml).
End diastolic volume | 12 months
  Echocardiogram assessment on volume of blood in the left ventricle at the end of diastolic filling (cc)
Left ventricular ejection fraction (LVEF) | 12 months
  Calculated by dividing the volume of blood pumped from the left ventricle per beat (stroke volume) by the volume of blood collected in the left ventricle at the end of diastolic filling (end-diastolic volume).
Participants Functional Activity by NYHA Classification | 12 months
  The New York Heart Association (NYHA) Functional Classification is a useful tool for classifying the extent of functional limitations in patients with heart conditions. The system categorizes patients into one of four categories based on the level of limitation they experience during physical activity, with symptoms ranging from mild shortness of breath or angina to more severe breathing difficulties. The NYHA classification focuses specifically on limitations related to physical activity and provides a straightforward approach to assessing a patient's condition. By using this system, healthcare providers can quickly and easily determine the level of functional limitation in their patients and tailor treatment plans accordingly.
Participants Functional Activity by CCS Classification | 12 months
  The Canadian Cardiovascular Society grading of angina pectoris, also known as the CCS Functional Classification, is a widely used clinical tool that classifies the severity of exertional angina. It allows doctors to assess the degree of angina severity in patients, and subsequently develop a tailored treatment plan. Although there are no definitive therapy guidelines specific to each class, healthcare providers can use the CCS grading system as a framework to guide treatment planning based on the severity of angina and other individual factors such as age and the risk of major cardiac complications. By utilizing the CCS grading system, healthcare providers can ensure that patients receive personalized treatment that addresses their unique needs and circumstances.

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - Chung Shan Medical University Hospital, Taichung, Taichung City
  - HONYA Medical Inc, Tainan

IPD SHARING:
Plan to Share IPD: No